CLINICAL TRIAL: NCT05068440
Title: A Phase 2, Single-Arm, Open-Label, Multicenter Study of the Bruton Tyrosine Kinase Inhibitor Zanubrutinib in Patients With CD79B Mutant Relapsed/Refractory Diffuse Large B-Cell Lymphoma
Brief Title: Treatment of CD79B Mutant Relapsed/Refractory Diffuse Large B-Cell Lymphoma With Bruton Tyrosine Kinase Inhibitor Zanubrutinib
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: BeiGene (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BGB-3111-218; CTR20210786 (Registry Identifier: ChinaDrugTrials)
Record Dates: First submitted 2021-09-27; First posted 2021-10-05 (Actual); Last update posted 2025-07-25 (Actual); Status verified 2025-07

CONDITIONS: Relapsed Diffuse Large B-cell Lymphoma; Refractory Diffuse Large B-cell Lymphoma
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse | interventions — zanubrutinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Zanubrutinib (Experimental): administered orally
  Interventions: Drug: Zanubrutinib

INTERVENTIONS:
Drug: Zanubrutinib — administered orally as capsules
  Other Names: BGB-3111; Brukinsa

SUMMARY:
Study consists of a single arm to explore the efficacy and safety of zanubrutinib in participants with CD79B mutant Relapsed/Refractory Diffuse Large B-Cell Lymphoma.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed DLBCL based on the World Health Organization (WHO) 2008 classification of tumors of hematopoietic and lymphoid tissue.
2. Positive CD79B mutation confirmed by the central laboratory.
3. Previously received at least 1 line of adequate systemic anti-DLBCL therapy, defined as an anti-CD20 antibody-based chemoimmunotherapy for at least 2 consecutive cycles, unless participants had disease progression before Cycle 2
4. Relapsed or refractory (R/R) disease before study entry, defined as either

   1. Recurrent disease after having achieved disease remission (CR or partial response [PR]) at the completion of the latest treatment regimen.
   2. Stable disease or PD at the completion of the latest treatment regimen
5. Ineligible for high dose therapy/stem cell transplantation, which is defined as meeting any of the following criteria:

   1. Significant organ dysfunction (eg, left ventricular ejection fraction < 50% by echocardiogram or multiple gated acquisition scan [MUGA], diffuse lung capacity for carbon monoxide < 60% predicted by pulmonary function test, creatinine clearance < 70 mL/min shown by nuclear medicine scan or 24-hour urine collection) or comorbidities precluding the use of high dose therapy/stem cell transplantation on the basis of unacceptable risk of treatment-related morbidity
   2. Failure to achieve CR or PR with salvage therapy.
   3. Failure to collect stem cells or unable to perform stem cell collection as assessed by the investigator.

Exclusion Criteria:

1. Participants who have NHL other than classical histology DLBCL (DLBCL, not otherwise specified), eg, participants with DLBCL transformed from indolent lymphomas, primary mediastinal (thymic) large B-cell lymphoma, primary cutaneous DLBCL, primary effusion lymphoma, and central nervous system (CNS) lymphoma.
2. History of allogeneic stem cell transplantation or chimeric antigen receptor (CAR) T-cell therapy.
3. Prior exposure to a Bruton's tyrosine kinase (BTK) inhibitor.
4. Receipt of the following treatment at the time indicated before the first dose of study drug:

   1. Corticosteroid given with antineoplastic intent within 2 weeks, but a short course (≤ 7 days) of systemic corticosteroid treatment at doses ≤ 20 mg/day prednisone equivalent for control of lymphoma-related symptoms is allowed prior to enrollment provided that it is tapered off within 5 days after initiation of study treatment.
   2. Chemotherapy or radiotherapy within 2 weeks.
   3. Monoclonal antibody within 2 weeks.
   4. Investigational therapy within 2 weeks.
   5. Chinese patent medicine with antineoplastic intent within 2 weeks.
5. History of other active malignancies within 2 years before study entry, with the exception of (1) adequately treated in-situ carcinoma of the cervix; (2) localized basal cell or squamous cell carcinoma of the skin; (3) previous malignancy confined and treated locally (surgery or other modality) with curative intent.

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2021-08-11 (Actual); Primary Completion 2025-03-31 (Actual); Study Completion 2025-03-31 (Actual)

PRIMARY OUTCOMES:
Overall response rate (ORR) | approximately 2 years
  Defined as the proportion of participants who achieved complete response (CR) or partial response (PR) by investigator assessment according to the Lugano classification for Non-Hodgkin's Lymphoma (NHL).

SECONDARY OUTCOMES:
Overall response rate (ORR) | approximately 3.5 years
  Defined as the proportion of participants who achieved complete response (CR) or partial response (PR) by Independent Review Committee assessment according to the Lugano classification for Non-Hodgkin's Lymphoma (NHL).
Complete response rate (CRR) | approximately 3.5 years
  Defined as the proportion of participants with a documented CR determined by the Independent Review Committee and by investigator assessment
Duration of response (DOR) | approximately 3.5 years
  DOR is defined as the time from the date of the first documented response (PR or better) after treatment initiation until the date of first documented disease progression or death, whichever occurs first. Determined by the Independent Review Committee and by investigator assessment
Progression-free survival (PFS) | approximately 3.5 years
  PFS is defined as time from start of treatment to the first documentation of disease progression or death, whichever occurs first as determined by the Independent Review Committee and by investigator assessment
Time to response (TTR) | approximately 3.5 years
  TTR is defined as the time from start of treatment to first documentation of response of Partial Response (PR) or better as determined by the Independent Review Committee and by investigator assessment
Overall survival (OS) | approximately 3.5 years
  OS defined as the time from start of treatment to the date of death due to any cause
Number of participants with adverse events | approximately 3.5 years
  Number of participants with adverse events and serious adverse events, including clinical laboratory measurements, physical examination, and vital signs

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — BeiGene
Locations (25):
- China (25):
  - Anhui Provincial Cancer Hospital Aka West Branch of Anhui Province Hospital, Hefei, Anhui
  - Beijing Friendship Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Fujian Cancer Hospital, Fuzhou, Fujian
  - Sun Yat Sen University Cancer Center, Guangzhou, Guangdong
  - Guangdong Provincial Peoples Hospital Huifu Branch, Guangzhou, Guangdong
  - The First Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong
  - The First Affiliated Hospital of Shantou University Medical College, Shantou, Guangdong
  - Hainan Cancer Hospital, Haikou, Hainan
  - Harbin Medical University Cancer Hospital, Harbin, Heilongjiang
  - Henan Cancer Hospital, Zhengzhou, Henan
  - Union Hospital of Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei
  - Tongji Hospital of Tongji Medical College Huazhong University of Science and Technology, Wuhan, Hubei
  - The Second Xiangya Hospital of Central South University, Changsha, Hunan
  - Hunan Cancer Hospital, Changsha, Hunan
  - The First Affiliated Hospital of Nanchang University Branch Donghu, Nanchang, Jiangxi
  - The First Hospital of Jilin University, Changchun, Jilin
  - Liaoning Cancer Hospital and Institute, Shenyang, Liaoning
  - Rui Jin Hospital Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality
  - Shanxi Provincial Cancer Hospital, Taiyuan, Shanxi
  - West China Hospital, Sichuan University, Chengdu, Sichuan
  - Institute of Hematology and Hospital of Blood Disease, Tianjin, Tianjin Municipality
  - Yunnan Cancer Hospital, Kunming, Yunnan
  - The First Affiliated Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - Zhejiang University College of Medicine Second Affiliated Hospital, Hangzhou, Zhejiang
  - Taizhou Hospital of Zhejiang, Taizhou, Zhejiang

IPD SHARING:
Plan to Share IPD: Yes
BeiGene shares data on completed studies responsibly and provides qualified scientific and medical researchers access to data and supporting documentation for clinical trials in dossiers for medicines and indications after submission and approval in the United States, China, and Europe. Clinical trials supporting subsequent local approvals, new indications, or combination products are eligible for sharing once corresponding regulatory approvals are achieved.
  BeiGene shares data only when permitted by applicable data privacy and security laws and regulations, when it is feasible to do so without compromising the privacy of study participants, and other considerations.
  Qualified researchers with appropriate competencies who are engaged in novel scientific research may submit a request for participant-level data with a research proposal for BeiGene review. Research teams must include a biostatistician and sign a Data Sharing Agreement prior to receiving access to clinical trial data.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: See plan description
Access Criteria: See plan description
URL: https://beigene.com/science/clinical-trials/